CLINICAL TRIAL: NCT06979622
Title: Electromagnetic Positioning-Assisted Ultrasound Guidance in Transjugular Intrahepatic Portosystemic Shunt (TIPS): A Prospective, Single-Arm Study
Brief Title: Electromagnetic Positioning-Assisted Ultrasound Guidance in Transjugular Intrahepatic Portosystemic Shunt (TIPS)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2025-136
Record Dates: First submitted 2025-05-13; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Portal Hypertension
Keywords: TIPS; Electromagnetic; ultrasound
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TIPS procedure under ultrasound combined with electromagnetic positioning guidance (Experimental)
  Interventions: Other: ultrasound combined with electromagnetic positioning guidance

INTERVENTIONS:
Other: ultrasound combined with electromagnetic positioning guidance — TIPS procedure under ultrasound combined with electromagnetic positioning guidance

SUMMARY:
Transjugular intrahepatic portosystemic shunt (TIPS) is an important method for treating complications related to portal hypertension. The difficulty of its surgical procedures lies in portal vein puncture. Improper operation may lead to complications such as hepatic artery hemorrhage, hepatic capsular hemorrhage, and biliary tract hemorrhage. At present, the means of guiding portal vein puncture are limited. There is evidence supporting that ultrasound guidance can help reduce the number of punctures and lower the radiation dose, etc. However, ordinary ultrasound is limited by the influence of dimensions and can only guide punctures in the same plane, with limited guiding value. The use of the Imedis9000 magnetic navigation system can guide percutaneous vascular puncture in multiple dimensions, which can increase the success rate of puncture and shorten the operation time. This study conducted a prospective, single-arm study. The Imedis9000 magnetic navigation system was used for real-time positioning to guide precise TIPS stent implantation. The number of punctures, puncture success rate, stent implantation success rate, and the incidence of adverse events were evaluated to determine the application value of the Imedis9000 magnetic navigation system in TIPS procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years old;
* Including but not limited to patients requiring TIPS for: acute esophageal/gastric variceal bleeding, portal hypertensive gastropathy, cirrhotic ascites, cirrhotic hydrothorax, hepatorenal syndrome, Budd-Chiari syndrome, atypical portal hypertension, portal vein thrombosis, prevention of recurrent esophageal/gastric variceal bleeding, or prevention of recurrent ectopic variceal bleeding;
* Deemed by clinicians to require Transjugular Intrahepatic Portosystemic Shunt (TIPS)
* Voluntarily signed informed consent form

Exclusion Criteria:

* Severe right heart failure, congestive heart failure (ejection fraction <40%), or severe valvular heart disease;
* Persistent severe pulmonary hypertension (mean pulmonary artery pressure >45 mmHg) despite treatment;
* Uncontrolled systemic infection or inflammation;
* Hepatic encephalopathy stage III-IV;
* Presence of cardiac pacemaker, metallic implants, or other conditions susceptible to electromagnetic interference;
* Pregnancy or lactation;
* Poor visualization of the portal venous system on ultrasound;
* Investigator-determined unsuitability for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2025-05-31 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Success rate of portal vein puncture | During TIPS procedure
  Puncture success rate = Number of successful cases/total number of cases ×100%.

IPD SHARING:
Plan to Share IPD: Undecided